CLINICAL TRIAL: NCT05280938
Title: A Randomized Clinical Trial on Mindfulness for African American Mothers Postpartum
Brief Title: Mindfulness for African Americans Postpartum
Acronym: MAAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, lgarfield, Assistant Professor, Loyola University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 212354; K23NR019101 (NIH)
Record Dates: First submitted 2022-02-24; First posted 2022-03-15 (Actual); Last update posted 2024-08-28 (Actual); Status verified 2024-08

CONDITIONS: Mental Disorders of Mother, Postpartum

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MAAP Intervention (Experimental): The MAAP intervention is an 8-week adapted mindfulness intervention based upon Kabat-Zinn's MBSR. The intervention includes spirituality, self-empowerment, interdependence, and story-telling which are salient to AAW. Session topics include Tasting Your Life, Seeing and Believing, The Scent of Roses, When Life Hurts, Hearing Your Own Cries, Embracing Inner Peace, Holding on, Welcoming Stillness. Each session will include an introduction, opening mindfulness practice, class responses to the previous week, review guidelines for class, guided individual reflection, group go-around/discussion, yoga, abdominal breathing, body scan, conclusion, and home practice. Face to face sessions 1, 4, 8 will be in a quiet room to allow group sitting or free floor space. Sessions 2, 3, 5, 6, are virtual on the zoom app. Participants receive practice links and a program workbook. Program attendance, type/amount of practice (weekly logs), and changes in mindfulness will be included in data analysis.
  Interventions: Behavioral: MAAP
- Educational Program (Active Comparator): The Education Program (attention control group) will be an 8-week educational program matched in duration and frequency to the MAAP intervention. Session topics are:1) Perineum and Incision Care, 2) Safe Sexual Practices, 3) Understanding Infant Feeding Methods, 4) How to Communicate Effectively with your Child's Health Care Providers, 5) Healthy Eating, 6) Infant Changing and Baths, 7) Infant Safety at Home, and 8) Utilizing Support from Family and the Community.
  Sessions will be given in groups by the same expert clinicians/educators for all cohorts. Subject receipt of the attention control will be monitored by attendance. Control group instructor will not include content on stress reduction or methods (yoga, meditation, etc.) taught in the MAAPI intervention. Classes will be given in the same setting as the MAAPI intervention, at the same time but on a different evening, to avoid crossover of effects.
  Interventions: Behavioral: Educational Program

INTERVENTIONS:
Behavioral: MAAP — Women randomized to the MAAP intervention will complete an 8 week (2hr/wk) hybrid adapted Kabat-Zinn's MBSR.(Kabat-Zinn, 1990) MAAP intervention includes activities related to spirituality, self-empowerment, interdependence, and story-telling, which are salient to AAW.(Watson-Singleton et al., 2019) Women will receive practice links and a program work book (5th grade level) containing objectives and weekly MAAP activities/. Individual weekly home practice is expected. Type and minutes of home practice will be recorded in weekly logs. Program attendance, type, amount of practice, and changes in mindfulness (Five Facet Mindfulness Questionnaire) will be included in data analysis.
  Arms: MAAP Intervention
Behavioral: Educational Program — The 8-week Educational Program will be matched in duration, frequency, delivery method, and data collection to the MAAP intervention. Like MAAP, it will be delivered using a hybrid format (virtual Zoom and in person visits).
  Sessions will be given in groups by an expert perinatal clinician/educator for all cohorts. Content will be "set" and delivered consistently across cohorts. Sessions will be audiotaped and rated for achievement of objectives and consistency of delivery. Deviations will be promptly addressed. Subject receipt will be monitored by attendance. Sessions will not include content on stress reduction (yoga, meditation, etc.). Classes will be given in the same setting as the MAAP intervention, at the same time but on a different evening, to avoid crossover (diffusion) of effects.
  Arms: Educational Program

SUMMARY:
A randomized clinical trial (RCT) design will be used to compare an 8-week Mindfulness for African Americans Postpartum (MAAP) intervention to an 8-week Educational Program (active comparison group). The primary objective is to evaluate the effectiveness of MAAP to decrease maternal psycho-behavioral symptoms and to improve mother/infant bonding. To better meet the needs of new mothers, MAAP will use a online form of delivery (i.e., group synchronous virtual Zoom). A secondary objective is to explore proinflammatory cytokines and oxytocin as possible biological mechanisms by which the MAAP intervention might decrease psycho-behavioral symptoms and improve mother/infant bonding. The MAAP intervention includes best approach and is culturally adapted based on prior evidence and expert opinion, and it addresses weaknesses in rigor of prior studies.

DETAILED DESCRIPTION:
This project is a first step to assess a culturally-tailored Mindfulness Intervention for African Americans Postpartum (MAAP). Elevated perinatal depressive symptoms are more common among disadvantaged African American women (AAW), 40-60%, compared to the national average,11-14 and AAW are almost four times as likely to have postpartum posttraumatic stress (13.4% vs 3.5%).15 Further, AAW are twice as likely to have a low birth weight infant (13.2% vs. 7%)16 and 1.6 times more likely to deliver preterm (16.3% vs. 10.2%) compared to non-Hispanic White women.17 AAW with preterm/low birthweight infants are at increased risk for psycho-behavioral disturbances and related impairments of infant development. This is a critical public health disparity.

The MAAP intervention is culturally adapted for AAW and includes using an AAW interventionist, providing course material that use written and artistic expressions of AAW with illustrations that portray AAW, creation of a community among research participants, inclusion of self-empowerment strategies, and the use of storytelling that resonates with AAW experience. The Investigators propose a randomized clinical trial to test the MAAP intervention compared to an Educational Program. This study aims to determine the extent to which MAAP affects psycho-behavioral symptoms and evaluate the effects of MAAP on pro- and anti-inflammatory biomarkers (proinflammatory cytokines and oxytocin). The Investigators will measure stress, depressive symptoms, anxiety, poor sleep, posttraumatic stress, fatigue, pro-inflammatory cytokines, and oxytocin to determine relationships among these variables and the MAAP intervention versus the Educational Program. The Investigators hypothesize participants in the MAAP intervention will have greater improvement of psycho-behavioral symptoms compared to participants in the Educational Program. The Investigators also hypothesize women in the MAAP intervention will have a greater decrease in pro-inflammatory cytokines and a greater increase in oxytocin compared to the Educational Program. The findings of this study will lay the groundwork for future research by identifying best-practice recruitment strategies, refining measurement strategies, and evaluating feasibility and acceptability.

A member of the research team, NICU nurses, and physicians will identify eligible subjects by daily unit census report. Multiple culturally competent strategies will be used to maximize subject recruitment and retention of AAW. The Investigators will be using an AAW interventionist, providing course material that use written and artistic expressions of AAW with illustrations that portray AAW, creation of a community among research participants, inclusion of self-empowerment strategies, and the use of storytelling that resonates with AAW experience. For recruitment, a NICU healthcare provider will make the first contact with a potential participant and then the PI or perinatal research assistant will further explain the study and informed consent. After informed consent, women will be randomized. The biostatistician will prepare sealed envelopes, using a block size of 4 participants. The MAAPI intervention and the Educational Program have a fixed time of 8 weeks, and will be run continuously allowing for 6 start times per year. Eight weeks will also serve as the recruitment time frame per cohort, estimating cohort size between 3-5 participants per group. Data will be collected at 3 times for both groups: T1=1st week session; T2= 4th week session; T3 = 8th week (conclusion). T1 will correspond to the first face to face meeting of the MAAP intervention or Educational Program. T1 data will be collected at the beginning of week 1 procedures for both the MAAP group and the Educational Program group. The Investigators estimate an ample recruitment window of 2 months per group will allow assembly of a cohort of at least three participants per group. using this design, the range of time elapsed from birth to a woman's entry into the intervention will vary and will be controlled in the statistical analysis.

Women randomized to the MAAP intervention will complete an 8 week (2hr/wk) hybrid adapted Kabat- Zinn's MBSR. MAAP intervention includes activities related to spirituality, self-empowerment, interdependence, and story-telling, which are salient to AAW. Session topics include 1) Tasting your Life, 2) Seeing and Believing, 3) The scent of Roses, 4) When Life Hurts, 5) Hearing Your Own Cries, 6) Embracing Inner Peace, 7) Holding On, 8) Welcoming Stillness. A manual has been developed for the MAAPI intervention with detailed protocols for each session. Face to face sessions (weeks 1, 4, and8) will be in a quiet room with movable chairs to allow group sitting or free floor space. Sessions for weeks 2, 3, 5, 6, 7 will be virtual classes offered via Zoom. Women will receive practice links and a program work book (5th grade level) containing objectives and weekly MAAP activities. Individual weekly home practice is expected. Type and minutes of home practice will be recorded in weekly logs. Program attendance, type, amount of practice, and changes in mindfulness (Five Facet Mindfulness Questionnaire) will be included in data analysis.

Participants randomized to the Educational Program will complete an 8 week (2hr/wk) hybrid educational program matched in duration, frequency, delivery method, and data collection to the MAAP intervention.Like MAAP, it will be delivered using a hybrid format (virtual Zoom and face-to-face sessions). Face-to-face sessions (weeks 1, 4, & 8) will be in a quiet room with movable chairs to allow group sitting or free floor space. Sessions for weeks 2, 3, 5, 6, 7 will be virtual classes offered via Zoom. At session week 1, participants will set up the Zoom app to ensure capabilities. Session topics are: 1) Perineum and Incision Care, 2) Safe Sexual Practices, 3) Understanding Infant Feeding Methods, 4) How to communicate Effectively with your Child's Health Care Providers, 5) Healthy Eating, 6) Infant Changing and Baths, 7) Infant Safety at Home, and 8) Utilizing Support from Family and the Community. Program content and objectives were reviewed by content experts (Neonatal Nurse Practitioner and Women's Health Nurse Practitioner. Sessions will be given in groups by an African American expert perinatal clinician/educator (not the PI) for all cohorts. Fidelity will be similar to that described for the MAAP intervention. Content will be "set" and delivered consistently across cohorts. Subject receipt will be monitored by attendance. Sessions will not include content on stress reduction (yoga, meditation, etc). Classes will be given in the same setting as the MAAP intervention, at the same time but on a different evening, to avoid crossover (diffusion) of effects.

The Investigators will use strategies to maximize retention and decrease missing data. These strategies include: 1) Establish project identity to increase subject engagement with the study. 2) Provide phone calls and texts one day prior to weekly session; on-going contacts with subjects. 3) Train nurse research assistants in subject retention strategies and subject follow-up. 4) Women who miss a session (face to face or virtual) will be telephoned to determine reason for absence and address any concerns that may inhibit participation in the project. If the Investigators are unable to reach participants by phone, the Investigators will leave a letter by the infant bedside, and mail a letter to her home address. Participants whose infants have been discharged will have the option of bringing their infants to the face to face sessions and scheduling home visits for data collection of saliva samples and questionnaires at T1, T2, and T3. Recruitment and retention progress and issues will be addressed with the study Mentoring Team and the Data Safety Monitoring Board. Multiple culturally adapted strategies will be used to maximize subject recruitment and retention of AAW. These include mindfulness sessions incorporating the concepts of spirituality, self-empowerment, and interdependence. The MAAP interventionist and the Research Assistant running the Educational Program will both identify as single or multiracial African American or black. Additionally, the MAAP workbook is specific to AAW, including writings and artistic expressions by AAW, and use of images of AAW in meditation/yoga poses. Our research plan already uses some of the recommended recruitment and retention strategies (i.e., compensation and consideration of personal or family medical problem).

The study was designed to enroll 40 participants, 20 in the MAAP intervention and 20 in the Education Program. The sample size of 40 was computed based on our primary hypothesis, that the MAAP intervention will have a greater improvement of psycho-behavioral symptoms, decreased pro-inflammatory cytokines, and increased oxytocin in African American women with a preterm/low birthweight infant compared to the Educational Program. Based on our pilot and published data, the effect size was estimated at 0.70 for anxiety, 0.45 for prenatal stress and 0.8 for sleep quality, 0.40 for depressive symptoms and 0.36 for proinflammatory cytokines. A sample size of 40 will achieve 80% power, given current effect size estimates per aim. To determine the extent to which the MAAP intervention improves maternal psycho-behavioral symptoms the Investigators will use growth curve analysis (HLM). HLM model longitudinal data by allowing random effects to account for repeated measures on participants over 3 times, and to evaluate change in trajectories over time. HLMs allow for analysis of unbalanced data across time points, increasing power and reducing bias. HLM analysis will evaluate the effects of the MAAP intervention on change in proinflammatory cytokines and oxytocin levels. Models will control for maternal age and gestational age at delivery.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible to participate in this study, an individual must meet all of the following criteria.

1. Participants must identify as African American/Black and have given birth to an infant
2. Participants will be over the age of 18 and able to speak and read English at a 5th grade level or above.
3. Participants must be willing to comply with study procedures including completion of an 8-week intervention or educational program, provide saliva samples 3 times at session 1, 4, and 8, answer questionnaires concerning demographics, and psycho-behavioral health symptoms, and be available for in person and virtual sessions during the duration of the study.
4. Participants must be willing to adhere to the MAAP intervention.
5. Participants must have access to a smart phone and agree to download the free app Zoom
6. Participants must sign and date an informed consent document -

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation:

1. Participants will be excluded from the study if they are currently using immune medications such as steroids, whether prescribed or not
2. Participants are excluded from the study if they have a diagnosis or disease process (physical or psychological) that precludes participation in the MAAP intervention.

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2022-02-07 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Parental Stress Level | Baseline (week 1)
  Stress is this proposal specifically measures how a participant feels regarding her infant. Stress will be measured with the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS: NICU). PSS: NICU has good construct validity and uses 28 items, rated on a 5-point Likert scale. Maternal perceived stress is measured using 3 sub-scales: 1) Stress experienced by parents from appearance, 2) behavior of their child, 3) the NICU environment affecting parenting role. Cronbach's alphas for the sub-scales are reported to be .80-.87, and the Cronbach's alpha is .88 for the total scale. This instrument is specifically tailored to parents with infants in the NICU and questions include: How stressful it is to see your infant with tubes or other devices, How stressful it is to witness your infant's behavior such as breathing difficulty, and How stressful it is to be a parent and not able to fully are for your infant.
Parental Stress Level | mid treatment (week 4)
  Stress is this proposal specifically measures how a participant feels regarding her infant. Stress will be measured with the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS: NICU). PSS: NICU has good construct validity and uses 28 items, rated on a 5-point Likert scale. Maternal perceived stress is measured using 3 sub-scales: 1) Stress experienced by parents from appearance, 2) behavior of their child, 3) the NICU environment affecting parenting role. Cronbach's alphas for the sub-scales are reported to be .80-.87, and the Cronbach's alpha is .88 for the total scale. This instrument is specifically tailored to parents with infants in the NICU and questions include: How stressful it is to see your infant with tubes or other devices, How stressful it is to witness your infant's behavior such as breathing difficulty, and How stressful it is to be a parent and not able to fully are for your infant.
Parental Stress Level | end of treatment (week 8)
  Stress is this proposal specifically measures how a participant feels regarding her infant. Stress will be measured with the Parental Stressor Scale: Neonatal Intensive Care Unit (PSS: NICU). PSS: NICU has good construct validity and uses 28 items, rated on a 5-point Likert scale. Maternal perceived stress is measured using 3 sub-scales: 1) Stress experienced by parents from appearance, 2) behavior of their child, 3) the NICU environment affecting parenting role. Cronbach's alphas for the sub-scales are reported to be .80-.87, and the Cronbach's alpha is .88 for the total scale. This instrument is specifically tailored to parents with infants in the NICU and questions include: How stressful it is to see your infant with tubes or other devices, How stressful it is to witness your infant's behavior such as breathing difficulty, and How stressful it is to be a parent and not able to fully are for your infant.
Depressive Symptoms | Baseline (week 1)
  Depressive symptoms include feelings of sadness and loss of interest and can affect sleep, eating, anxiety, trouble concentrating, self-blame, and unexplained physical discomfort. These symptoms can cause difficulty with day to day activities including difficulty with maternal interactions with her infant and daily infant care. Postpartum depressive symptoms are depressive symptoms occurring during the postpartum time which has been defined as up to 4 weeks postpartum ranging to up to one year postpartum. Depressive symptoms will be measured with the Center for Epidemiologic Studies Depression Scale (CESD). The CESD is a self-report measure consisting of 20 depressive symptoms items and rated on a 4-point Likert Scale. Scores range from 0-60. Higher scores indicate more depressive symptoms. Scores >15 indicate elevated depressive symptoms. Cronbach's alpha = .87-91 in minority mothers of preterm infants.
Depressive Symptoms | mid treatment (week 4)
  Depressive symptoms include feelings of sadness and loss of interest and can affect sleep, eating, anxiety, trouble concentrating, self-blame, and unexplained physical discomfort. These symptoms can cause difficulty with day to day activities including difficulty with maternal interactions with her infant and daily infant care. Postpartum depressive symptoms are depressive symptoms occurring during the postpartum time which has been defined as up to 4 weeks postpartum ranging to up to one year postpartum. Depressive symptoms will be measured with the Center for Epidemiologic Studies Depression Scale (CESD). The CESD is a self-report measure consisting of 20 depressive symptoms items and rated on a 4-point Likert Scale. Scores range from 0-60. Higher scores indicate more depressive symptoms. Scores >15 indicate elevated depressive symptoms. Cronbach's alpha = .87-91 in minority mothers of preterm infants.
Depressive Symptoms | end of treatment (week 8)
  Depressive symptoms include feelings of sadness and loss of interest and can affect sleep, eating, anxiety, trouble concentrating, self-blame, and unexplained physical discomfort. These symptoms can cause difficulty with day to day activities including difficulty with maternal interactions with her infant and daily infant care. Postpartum depressive symptoms are depressive symptoms occurring during the postpartum time which has been defined as up to 4 weeks postpartum ranging to up to one year postpartum. Depressive symptoms will be measured with the Center for Epidemiologic Studies Depression Scale (CESD). The CESD is a self-report measure consisting of 20 depressive symptoms items and rated on a 4-point Likert Scale. Scores range from 0-60. Higher scores indicate more depressive symptoms. Scores >15 indicate elevated depressive symptoms. Cronbach's alpha = .87-91 in minority mothers of preterm infants.
Anxiety Level | Baseline (week 1)
  Anxiety includes feelings of worry, nervousness, fear, unease, or excess uncertainty. State anxiety is a transient reaction directly related to an adverse situation and will be measured in this proposal. Maternal state anxiety will be measured with the state anxiety sub-scale of the State-Trait Anxiety Inventory (STAI). The state sub-scale consists of 20 items rated on a 4-point Likert scale and includes topics such as the degree to which the mother currently feels happy, calm, comfortable, jittery, upset, and confused. A higher score is associated with higher levels of anxiety. Cronbach's alphas .85-.95. Numerous reliability and validity studies of the STAI have been conducted with coefficients ranging from .16-.53, as would be expected, as the STAI is designed to be influenced by situational factors.
Anxiety Level | mid treatment (week 4)
  Anxiety includes feelings of worry, nervousness, fear, unease, or excess uncertainty. State anxiety is a transient reaction directly related to an adverse situation and will be measured in this proposal. Maternal state anxiety will be measured with the state anxiety sub-scale of the State-Trait Anxiety Inventory (STAI). The state sub-scale consists of 20 items rated on a 4-point Likert scale and includes topics such as the degree to which the mother currently feels happy, calm, comfortable, jittery, upset, and confused. A higher score is associated with higher levels of anxiety. Cronbach's alphas .85-.95. Numerous reliability and validity studies of the STAI have been conducted with coefficients ranging from .16-.53, as would be expected, as the STAI is designed to be influenced by situational factors.
Anxiety Level | end of treatment (week 8)
  Anxiety includes feelings of worry, nervousness, fear, unease, or excess uncertainty. State anxiety is a transient reaction directly related to an adverse situation and will be measured in this proposal. Maternal state anxiety will be measured with the state anxiety sub-scale of the State-Trait Anxiety Inventory (STAI). The state sub-scale consists of 20 items rated on a 4-point Likert scale and includes topics such as the degree to which the mother currently feels happy, calm, comfortable, jittery, upset, and confused. A higher score is associated with higher levels of anxiety. Cronbach's alphas .85-.95. Numerous reliability and validity studies of the STAI have been conducted with coefficients ranging from .16-.53, as would be expected, as the STAI is designed to be influenced by situational factors.
Elevated Posttraumatic stress | Baseline (week 1)
  Postpartum post-traumatic stress is a type of stress affecting persons exposed to traumatic events. Elevated post-traumatic stress symptoms include 1) re-experiencing the event through thoughts, 2) avoidance of stimuli related to the event, and 3) increased arousal since the event. Post-traumatic stress symptoms after childbirth may be related to a traumatic childbirth experience or to a previous traumatic event in the mother's life. The Perinatal PTSD Questionnaire (PPQ) will measure the extent to which mothers experience post-traumatic stress symptoms in response to their birth experience. PPQ has 14 yes-no items that measure intrusive thoughts (e.g., bad dreams of giving birth), avoidance or numbing (e.g., inability to remember parts of the hospitalization), and increased arousal (e.g., increased irritability or anger). The "yes" answers are summed. Cronbach's alpha was .83 and test-retest reliability from 2 to 4 weeks was .92
Elevated Posttraumatic stress | mid treatment (week 4)
  Postpartum post-traumatic stress is a type of stress affecting persons exposed to traumatic events. Elevated post-traumatic stress symptoms include 1) re-experiencing the event through thoughts, 2) avoidance of stimuli related to the event, and 3) increased arousal since the event. Post-traumatic stress symptoms after childbirth may be related to a traumatic childbirth experience or to a previous traumatic event in the mother's life. The Perinatal PTSD Questionnaire (PPQ) will measure the extent to which mothers experience post-traumatic stress symptoms in response to their birth experience. PPQ has 14 yes-no items that measure intrusive thoughts (e.g., bad dreams of giving birth), avoidance or numbing (e.g., inability to remember parts of the hospitalization), and increased arousal (e.g., increased irritability or anger). The "yes" answers are summed. Cronbach's alpha was .83 and test-retest reliability from 2 to 4 weeks was .92
Elevated Posttraumatic stress | end of treatment (week 8)
  Postpartum post-traumatic stress is a type of stress affecting persons exposed to traumatic events. Elevated post-traumatic stress symptoms include 1) re-experiencing the event through thoughts, 2) avoidance of stimuli related to the event, and 3) increased arousal since the event. Post-traumatic stress symptoms after childbirth may be related to a traumatic childbirth experience or to a previous traumatic event in the mother's life. The Perinatal PTSD Questionnaire (PPQ) will measure the extent to which mothers experience post-traumatic stress symptoms in response to their birth experience. PPQ has 14 yes-no items that measure intrusive thoughts (e.g., bad dreams of giving birth), avoidance or numbing (e.g., inability to remember parts of the hospitalization), and increased arousal (e.g., increased irritability or anger). The "yes" answers are summed. Cronbach's alpha was .83 and test-retest reliability from 2 to 4 weeks was .92
Sleep Quality | Baseline (week 1)
  Sleep disturbance includes difficulties falling asleep, staying asleep, and contributes to disease, impaired cognition, and poor quality of life. Sleep disturbances have been reported by many postpartum women and are associate with psycho-behavioral disturbances such as depressive symptoms. Maternal sleep quality will be measured by the Pittsburgh Sleep Quality Inventory (PSQI). The PSQI is a 19 question self-rated questionnaire which assesses sleep quality, has a global score of 0-21, and has 7 sub-scales. Higher scores indicate worse sleep quality. A PSQI score >5 yielded a sensitivity of 89.6% and a specificity of 86.5% in distinguishing good and poor sleepers. Internal consistency is .76-.83 and in perinatal women Cronbach's alpha ranges are .72-.78.
Sleep Quality | mid treatment (week 4)
  Sleep disturbance includes difficulties falling asleep, staying asleep, and contributes to disease, impaired cognition, and poor quality of life. Sleep disturbances have been reported by many postpartum women and are associate with psycho-behavioral disturbances such as depressive symptoms. Maternal sleep quality will be measured by the Pittsburgh Sleep Quality Inventory (PSQI). The PSQI is a 19 question self-rated questionnaire which assesses sleep quality, has a global score of 0-21, and has 7 sub-scales. Higher scores indicate worse sleep quality. A PSQI score >5 yielded a sensitivity of 89.6% and a specificity of 86.5% in distinguishing good and poor sleepers. Internal consistency is .76-.83 and in perinatal women Cronbach's alpha ranges are .72-.78.
Sleep Quality | end of treatment (week 8)
  Sleep disturbance includes difficulties falling asleep, staying asleep, and contributes to disease, impaired cognition, and poor quality of life. Sleep disturbances have been reported by many postpartum women and are associate with psycho-behavioral disturbances such as depressive symptoms. Maternal sleep quality will be measured by the Pittsburgh Sleep Quality Inventory (PSQI). The PSQI is a 19 question self-rated questionnaire which assesses sleep quality, has a global score of 0-21, and has 7 sub-scales. Higher scores indicate worse sleep quality. A PSQI score >5 yielded a sensitivity of 89.6% and a specificity of 86.5% in distinguishing good and poor sleepers. Internal consistency is .76-.83 and in perinatal women Cronbach's alpha ranges are .72-.78.
Fatigue Symptoms | Baseline (week 1)
  Fatigue is extreme tiredness resulting from mental or physical exertion. Symptoms of fatigue include tiredness, headache, aching/sore muscles, impaired decision-making and judgement, moodiness, and irritability. Fatigue has been reported in many postpartum women and is associate with psycho-behavioral disturbances. Maternal fatigue will be measured by the Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF). MFSI-SF is a 14 item self-report instrument that measure severity, frequency, and patterns of fatigue. The MFSI provides a score for overall fatigue in 5 domains (general, emotional, physical, mental, vigor). Factor analysis shows good fit and internal consistency ranges from .87-.96
Fatigue Symptoms | mid treatment (week 4)
  Fatigue is extreme tiredness resulting from mental or physical exertion. Symptoms of fatigue include tiredness, headache, aching/sore muscles, impaired decision-making and judgement, moodiness, and irritability. Fatigue has been reported in many postpartum women and is associate with psycho-behavioral disturbances. Maternal fatigue will be measured by the Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF). MFSI-SF is a 14 item self-report instrument that measure severity, frequency, and patterns of fatigue. The MFSI provides a score for overall fatigue in 5 domains (general, emotional, physical, mental, vigor). Factor analysis shows good fit and internal consistency ranges from .87-.96
Fatigue Symptoms | end of treatment (week 8)
  Fatigue is extreme tiredness resulting from mental or physical exertion. Symptoms of fatigue include tiredness, headache, aching/sore muscles, impaired decision-making and judgement, moodiness, and irritability. Fatigue has been reported in many postpartum women and is associate with psycho-behavioral disturbances. Maternal fatigue will be measured by the Multidimensional Fatigue Symptom Inventory Short Form (MFSI-SF). MFSI-SF is a 14 item self-report instrument that measure severity, frequency, and patterns of fatigue. The MFSI provides a score for overall fatigue in 5 domains (general, emotional, physical, mental, vigor). Factor analysis shows good fit and internal consistency ranges from .87-.96
Mindfulness | Baseline (week 1)
  Mindfulness is a mental state of focusing one's awareness on the present moment, acknowledging/accepting one's mental feelings, physical feelings, and thoughts. The Five Facets of Mindfulness Questionnaire (FFMQ) will be used to assess mindfulness. These facets include: observing,describing, acting with awareness, non-judging of inner experience, non-reactivity to inner experience. The FFMQ utility with African American samples is established with an internal consistency range of .60-.86
Mindfulness | mid treatment (week 4)
  Mindfulness is a mental state of focusing one's awareness on the present moment, acknowledging/accepting one's mental feelings, physical feelings, and thoughts. The Five Facets of Mindfulness Questionnaire (FFMQ) will be used to assess mindfulness. These facets include: observing,describing, acting with awareness, non-judging of inner experience, non-reactivity to inner experience. The FFMQ utility with African American samples is established with an internal consistency range of .60-.86
Mindfulness | end of treatment (week 8)
  Mindfulness is a mental state of focusing one's awareness on the present moment, acknowledging/accepting one's mental feelings, physical feelings, and thoughts. The Five Facets of Mindfulness Questionnaire (FFMQ) will be used to assess mindfulness. These facets include: observing,describing, acting with awareness, non-judging of inner experience, non-reactivity to inner experience. The FFMQ utility with African American samples is established with an internal consistency range of .60-.86

SECONDARY OUTCOMES:
Pro-inflammatory cytokines | Baseline (week 1)
  Inflammatory theories posit that stressful experiences stimulate the release of pro-inflammatory cytokines, which signal the brain to engender depressive behaviors. Saliva cytokine changes occur during pregnancy to ensure fetal development and maternal health. Pro-inflammatory cytokines will be assessed through saliva levels. IL-6 and TNF-alpha will be measured via ELISA assay. Samples will be run in duplicate. Sensitivity is < 0.7 pg/ml for IL-6, and <3.9 pg/ml for TNF-alpha. Intra assay variability is <7%.
Pro-inflammatory cytokines | mid treatment (week 4)
  Inflammatory theories posit that stressful experiences stimulate the release of pro-inflammatory cytokines, which signal the brain to engender depressive behaviors. Saliva cytokine changes occur during pregnancy to ensure fetal development and maternal health. Pro-inflammatory cytokines will be assessed through saliva levels. IL-6 and TNF-alpha will be measured via ELISA assay. Samples will be run in duplicate. Sensitivity is < 0.7 pg/ml for IL-6, and <3.9 pg/ml for TNF-alpha. Intra assay variability is <7%.
Pro-inflammatory cytokines | end of treatment (week 8)
  Inflammatory theories posit that stressful experiences stimulate the release of pro-inflammatory cytokines, which signal the brain to engender depressive behaviors. Saliva cytokine changes occur during pregnancy to ensure fetal development and maternal health. Pro-inflammatory cytokines will be assessed through saliva levels. IL-6 and TNF-alpha will be measured via ELISA assay. Samples will be run in duplicate. Sensitivity is < 0.7 pg/ml for IL-6, and <3.9 pg/ml for TNF-alpha. Intra assay variability is <7%.
oxytocin | Baseline (week 1)
  Oxytocin is essential to the initiation of nurturing maternal behaviors and bonding between mother and child. Oxytocin release promotes actions relating to the development of social attachments. Low levels of oxytocin are linked to less touch between mothers and infants; whereas high levels of oxytocin are associated with increased gaze, vocalization, positive affect, and touch. Saliva oxytocin will be analyzed using an ELISA. Oxytocin detection levels are 15.6 pg/ml to 1000 pg/ml with sensitivity as low as 11.7 pg/ml. Intra-assay coefficient of variability range from 5-10% with an inter-assay coefficient of variability of 4.6% to 8.6%.
oxytocin | mid treatment (week 4)
  Oxytocin is essential to the initiation of nurturing maternal behaviors and bonding between mother and child. Oxytocin release promotes actions relating to the development of social attachments. Low levels of oxytocin are linked to less touch between mothers and infants; whereas high levels of oxytocin are associated with increased gaze, vocalization, positive affect, and touch. Saliva oxytocin will be analyzed using an ELISA. Oxytocin detection levels are 15.6 pg/ml to 1000 pg/ml with sensitivity as low as 11.7 pg/ml. Intra-assay coefficient of variability range from 5-10% with an inter-assay coefficient of variability of 4.6% to 8.6%.
oxytocin | end of treatment (week 8)
  Oxytocin is essential to the initiation of nurturing maternal behaviors and bonding between mother and child. Oxytocin release promotes actions relating to the development of social attachments. Low levels of oxytocin are linked to less touch between mothers and infants; whereas high levels of oxytocin are associated with increased gaze, vocalization, positive affect, and touch. Saliva oxytocin will be analyzed using an ELISA. Oxytocin detection levels are 15.6 pg/ml to 1000 pg/ml with sensitivity as low as 11.7 pg/ml. Intra-assay coefficient of variability range from 5-10% with an inter-assay coefficient of variability of 4.6% to 8.6%.

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Medical Center, Maywood, Illinois, United States

IPD SHARING:
Plan to Share IPD: No